CLINICAL TRIAL: NCT05854121
Title: Functional Electrical Stimulation Versus Constrained Induced Movement Therapy for Motor Recovery and Spasticity in Upper Limb Hemiparetic Chronic Ischemic Stroke Patients
Brief Title: FES VS Constrained Induced MT Recovery and Spasticity in Upper Limb Hemiparetic Ischemic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/531
Record Dates: First submitted 2023-03-18; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Electrical Stimulation (Other)
  Interventions: Diagnostic Test: Functional Electrical Stimulation
- Constrained Induced Movement Therapy (Experimental)
  Interventions: Diagnostic Test: Constrained Induced Movement Therapy

INTERVENTIONS:
Diagnostic Test: Functional Electrical Stimulation — Functional Electrical Stimulation for Motor Recovery and Spasticity in Upper Limb Hemiparetic Chronic Ischemic Stroke Patients
  Arms: Functional Electrical Stimulation
Diagnostic Test: Constrained Induced Movement Therapy — Constrained Induced Movement Therapy for Motor Recovery and Spasticity in Upper Limb Hemiparetic Chronic Ischemic Stroke Patients
  Arms: Constrained Induced Movement Therapy

SUMMARY:
To determines the effects of Functional Electrical Stimulation versus Constrained Induced Movement Therapy for motor recovery and spasticity in Upper Limb Hemiparetic Chronic Ischemic Stroke Patients

ELIGIBILITY:
Inclusion Criteria:

Clinically diagnosed chronic ischemic stroke patients. Patients from both genders Age 45 year and older. Patients having upper limb spasticity equal to 2 or less than 2 according to modified ash worth scale.

Patients having active cognitive scoring on Mini Mental State Examination.

Exclusion Criteria:

Having pacemaker and other stimulation devices. Prosthesis of bones, joints in targeted region of treatment. Patients presenting the history of recurrent stroke. Patients having history of bilateral hemiparesis. Co-morbid history of tumor, heart disease, hypertensive. Patients presenting with skin lesions, wounds, discoloration will be excluded from this research.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Scale Modified Ash worth | 6 Months
Motor Function assessment test | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Shadman Medical Care, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No